CLINICAL TRIAL: NCT03308617
Title: Sonication of Syndesmotic Screws
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jena University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: JenaUC
Record Dates: First submitted 2017-10-09; First posted 2017-10-12 (Actual); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Periimplant Infection
Keywords: sonication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — skin and wound swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Peri-implant infections are severe complications after internal fracture fixation surgery. Detection of causative agents of orthopedic implant-associated infections (OIAI) is demanding. Several authors reported increased identification rates of bacterial prevalence using different sonication procedures compared to standard tissue cultures samples, especially for low grade infections.

On the author hand, contamination of implants without clinical signs of infection is reported in up to 30% during implant removals after uneventful fracture healing. The raised general questions are: 1.) Is a positive microbiological finding the result of contamination during the index surgery or during implant removal? 2.) Does contaminated implants without clinical or serological signs of infection have a pathological value?

DETAILED DESCRIPTION:
In this prospective case study, the detection rates of different diagnostic tools for peri-implant contaminations during removal of syndesmotic screws should be compared and the clinical consequence of positive findings evaluated in follow up investigations up to 6 months.

Patients with ankle fractures (Weber B and C) treated operatively in our department by open reduction and internal fixation with plates and additional syndesmotic screw should be included. After patients´ informed consent, several microbiological samples should be taken for further microbiological analysis during the standard syndesmotic screw removal 6-8 weeks after the index surgery. At follow up of two weeks after screw removal a clinical examination and serological analysis for infection will be performed. The endpoint of study is fracture healing at six months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with syndesmotic screw removal after open reduction and internal fixation with plates and additional syndesmotic screw of ankle fractures (Weber B or C) in our department.

Exclusion Criteria:

* Patients with immunosuppressive diseases or therapies,
* Pregnant women
* Patients with pre-operations on the same ankle-joint
* Patients with initial surgery for fracture fixation in other hospitals.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with operatively treated ankle fractures.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Detection rate of syndesmotic screw contamination using a sonication procedure compared to standard wound swabs | six weeks

SECONDARY OUTCOMES:
Clinical manifestation of infections by contaminated fracture fixation implants | six months

CONTACTS AND LOCATIONS:
Overall Officials: Florian Gras, PD Dr. med., Principal Investigator — Department of Trauma-, Hand- and Reconstructive Surgery
Locations (1):
- Department of Trauma-, Hand- and Reconstructive Surgery, Jena, Thuringia, Germany

IPD SHARING:
Plan to Share IPD: No